CLINICAL TRIAL: NCT01433978
Title: A Phase 3, Multicenter, Randomized, Double-blind, Active-controlled, Parallel-group Trial With an Open-label Extension Phase to Evaluate the Efficacy and Safety of Oral E5501 Versus Eltrombopag, in Adults With Chronic Immune Thrombocytopenia (Idiopathic Thrombocytopenic Purpura)
Brief Title: A Phase 3, Multicenter, Randomized, Double-blind,Active-controlled, Parallel-group Trial With an Open-labelExtension Phase to Evaluate the Efficacy and Safety of OralE5501 Versus Eltrombopag, in Adults With Chronic ImmuneThrombocytopenia (Idiopathic Thrombocytopenic Purpura)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated early due to significant enrollment challenges.
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E5501-G000-305
Record Dates: First submitted 2011-09-13; First posted 2011-09-14 (Estimated); Results first posted 2018-02-06 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-01

CONDITIONS: Idiopathic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag; avatrombopag; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (3):
- Avatrombopag (Core Study) (Active Comparator): Avatrombopag will be administered orally as 5 mg, 10 mg, 20 mg, 30 mg or 40 mg in a flexible dose design for 26 weeks. Participants will receive blinded therapy at a starting dose of 20 mg avatrombopag, once daily and allow to have their dose titrated up (maximum dose of 40 mg avatrombopag) or down (minimum dose of 5 mg avatrombopag) depending on their response to study drug.
  Interventions: Drug: Avatrombopag; Drug: Standard of care
- Eltrombopag (Core Study) (Active Comparator): Eltrombopag will be administered orally as 25 mg, 50 mg, or 75 mg in a flexible dose design for 26 weeks. Participants will receive blinded therapy at a starting dose of 50 mg eltrombopag once daily and allow to have their dose titrated up (maximum dose of 75 mg eltrombopag) or down (minimum dose of 25 mg eltrombopag) depending on their response to study drug.
  Interventions: Drug: Eltrombopag; Drug: Standard of care
- Avatrombopag (Open-label Extension) (Experimental): Participants who meet the eligibility requirements for the Open-label Extension (OLE) Phase or who discontinue the Core Study early because of lack of treatment effect will be eligible to continue into the OLE Phase for up to 104 weeks of open-label avatrombopag therapy. Participants who enter the OLE from the Core Study will receive a starting dose of open-label avatrombopag which will be determined by the last dose of study drug at the End of Treatment (EOT) Visit (Visit 22) of the Core Study. Participants who discontinue the Core Study early because of lack of treatment effect and enter the OLE will receive open-label avatrombopag at a starting dose of 20 mg once daily of open-label avatrombopag.
  Interventions: Drug: Avatrombopag; Drug: Standard of care

INTERVENTIONS:
Drug: Eltrombopag
  Other Names: Promacta; Revolade
  Arms: Eltrombopag (Core Study)
Drug: Avatrombopag
  Other Names: E5501; Avatrombopag maleate
  Arms: Avatrombopag (Core Study); Avatrombopag (Open-label Extension)
Drug: Standard of care — Permitted ITP concomitant background therapies are as follows:
  * Corticosteroids and/or azathioprine taken at a stable dose for 4 weeks before randomization;
  * Mycophenolate mofetil (MMF) or danazol taken at a stable dose for at least 12 weeks before randomization;
  * Cyclosporine A (CsA) (due to the fact that it is a P-glycoprotein-mediated transport [P-gp] inhibitor) is to be avoided unless deemed medically necessary; CsA taken at a stable dose for at least 12 weeks before randomization.
  At the discretion of the investigator, participants will be allowed to use aspirin, other salicylates, or approved adenosine diphosphate (ADP) receptor antagonists, (eg, clopidogrel, prasugrel) during the study once their platelet count had risen.
  Participants treated with proton pump inhibitors (PPIs) and H2 antagonist therapy will receive a stable dose for at least 6 weeks prior to randomization. Treatment with these therapies must have been completed at least 2 weeks prior to randomization.

SUMMARY:
Core study:

To compare the efficacy of avatrombopag (in addition to standard) of care to eltrombopag (in addition to standard of care) for the treatment of adult participants with chronic immune thrombocytopenia (idiopathic thrombocytopenic purpura [ITP]) as measured by durable platelet response.

Open-label Extension Phase:

To evaluate the safety and tolerability of long-term therapy with avatrombopag in participants with chronic ITP (cITP).

DETAILED DESCRIPTION:
The study consists of three phases: Prerandomization, Randomization (Core Study) and Extension Phase. Participants 18 years of age and over, who meet all the eligibility requirements will be randomized into the study. It will require that splenectomized participants make up at least 35% of the study population and no single platelet count is greater than 35x10^9/L. Participants will be centrally stratified at randomization by splenectomy status, baseline platelet count, and use of concomitant ITP medication at baseline and randomized to receive either double-blind avatrombopag or eltrombopag in a 1:1 ratio. Participants will receive blinded therapy at a starting dose of 20 mg avatrombopag once daily or 50 mg eltrombopag once daily. Participants will be allowed to have their dose titrated up (maximum dose 40 mg avatrombopag and 75 mg for eltrombopag) or down (minimum dose 5 mg for avatrombopag and 25 mg for eltrombopag) depending on their response to study drug. The goal of dose modification is to maintain the platelet count at levels greater than or equal to 50x10^9/L and less than or equal to 150x10^9/L, and to decrease the need for ITP-directed concomitant medications. The duration of treatment in the Core study and the Extension Phase is approximately 26 and 104 weeks, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women greater than or equal to 18 years of age.
2. Participants diagnosed with cITP (greater than or equal to 12 months duration) according to the American Society for Hematology/British Committee for Standards in Hematology (ASH/BCSH) guidelines, and an average of 2 platelet counts less than 30x10^9/L). The physical exam should not suggest any disease which may cause thrombocytopenia other than ITP.
3. Participants who previously received one or more ITP therapies (including, but not limited to corticosteroids, immunoglobulins, azathioprine, danazol, cyclophosphamide and/or rituximab).
4. Participants must have had either initially responded (platelet count greater than 50x10^9/L) to a previous ITP therapy or have had a bone marrow examination consistent with ITP within 3 years to rule out myelodysplastic syndrome (MDS) or other causes of thrombocytopenia.
5. Prothrombin time/International Normalized Ratio (PT/INR) and activated partial thromboplastin time (aPTT) must have been within 80% to 120% of the normal range with no history of hypercoagulable state.
6. A complete blood count within the reference range (including white blood count [WBC] differential not indicative of a disorder other than ITP), with the following exceptions: a) Hemoglobin: participants with hemoglobin levels between 10 g/dL (100 g/L) and the lower limit of normal (LLN) are eligible for inclusion, if anemia was clearly attributable to ITP (excessive blood loss); b) Absolute neutrophil count (ANC) greater than or equal to 1500/uL (1.5x10^9/L) (elevated WBC/ANC due to corticosteroid treatment is acceptable).

Exclusion Criteria:

Core Study

1. Participants with known secondary immune thrombocytopenia (e.g., participants with known Helicobacter pylori-induced ITP, infected with known human immunodeficiency virus [HIV] or hepatitis C virus [HCV] or with known systemic lupus erythematosus [SLE]).
2. Participants considered unable, or unwilling to comply with the study protocol requirements or give informed consent, as determined by the investigator.
3. Participants with significant medical conditions that may impact the safety of the participant or interpretation of the study results (e.g., acute hepatitis, active chronic hepatitis; lymphoproliferative disease; myeloproliferative disorders, leukemia).
4. History of MDS.
5. History of pernicious anemia or participants with vitamin B12 deficiency who have not had pernicious anemia excluded as a cause.
6. Any prior history of arterial or venous thrombosis (stroke, transient ischemic attack, myocardial infarction, deep vein thrombosis, or pulmonary embolism), and more than two of the following risk factors: estrogen-containing hormone replacement or contraceptive therapies, smoking, diabetes, hypercholesterolemia, medication for hypertension, cancer, hereditary thrombophilic disorders (e.g., Factor V Leiden, antithrombin III deficiency, etc.), or any other family history of arterial or venous thrombosis.
7. Participants with a history of significant cardiovascular disease (e.g., congestive heart failure [CHF] New York Heart Association Grade III/IV), arrhythmia known to increase the risk of thromboembolic events [e.g., atrial fibrillation], participants with a QT interval corrected for heart rate of >450 msec, angina, unstable angina, coronary artery stent placement, angioplasty, or coronary artery bypass grafting).
8. Participants with a history of cirrhosis, portal hypertension, and chronic active hepatitis.
9. Participants with concurrent malignant disease.
10. Use of immunoglobulins (IVIg and anti-D) within 1 week of randomization.
11. Splenectomy or use of rituximab within 12 weeks of randomization.
12. Use of romiplostim or eltrombopag within 4 weeks of randomization.
13. Participants who are currently treated with corticosteroids or azathioprine but have not been receiving a stable dose for at least 4 weeks prior to randomization or have not completed these therapies more than 4 weeks prior to randomization.
14. Participants who are currently treated with MMF, CsA, or danazol but have not been receiving a stable dose for at least 12 weeks prior to randomization or have not completed these therapies more than 4 weeks prior to randomization.
15. Use of cyclophosphamide or vinca alkaloid regimens within 4 weeks of randomization.
16. Participants who are currently treated with PPIs or H2 antagonist therapy but have not been receiving a stable dose for at least 6 weeks prior to randomization or have not completed these therapies more than 2 weeks prior to randomization.
17. Fasting gastrin-17 blood levels exceeding ULN (including subjects on PPIs and H2 antagonists) at Screening.
18. Blood creatinine exceeding ULN by more than 20% OR total albumin below the LLN by 10% (revised per Amendment 01).
19. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels exceeding 2 times the ULN; total bilirubin exceeding 1.5 times the ULN.
20. Participants with a history of cancer treatment with cytotoxic chemotherapy and/or radiotherapy.
21. Participants with a history of ITP treatment with cytotoxic chemotherapy are still eligible for enrollment.
22. Females who are pregnant (positive beta-human chorionic gonadotropin [B-hCG] test) or breastfeeding.
23. Participants with a known allergy to E5501 or eltrombopag and any of their excipients.
24. Participants with a history of significant aminotransferase elevations while receiving eltrombopag (defined as ALT and/or AST elevation >3 x ULN).
25. Participants who are known nonresponders (defined as platelet counts that never exceed 50 x 10^9/L) to all previous TPO agonist therapy (including previous E5501 therapy) who do not have a bone marrow examination consistent with ITP taken at any point after failure of TPO therapy to rule out MDS or other causes of thrombocytopenia.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-03-26 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joe McIntosh, Study Director — Eisai Inc.
Locations (1):
- Prairie Lakes Health Care System, Watertown, South Dakota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One screen-failed participant was randomized into the study in error, but not dosed.
Groups:
- Eltrombopag (Core Study): Eltrombopag was administered orally as 25 mg, 50 mg, or 75 mg in a flexible dose design for 26 weeks. Participants received blinded therapy at a starting dose of 50 mg eltrombopag once daily and they were allowed to have their dose titrated up (maximum dose of 75 mg eltrombopag) or down (minimum dose of 25 mg eltrombopag) depending on their response to study drug.
- Avatrombopag (Core Study): Avatrombopag was administered orally as 5 mg, 10 mg, 20 mg, 30 mg or 40 mg in a flexible dose design for 26 weeks. Participants received blinded therapy at a starting dose of 20 mg avatrombopag, once daily and they were allowed to have their dose titrated up (maximum dose of 40 mg avatrombopag) or down (minimum dose of 5 mg avatrombopag) depending on their response to study drug.
- Avatrombopag (Open-label Extension Phase): Participants who met the eligibility requirements for the Open-label Extension (OLE) Phase or who discontinued the Core Study early because of lack of treatment effect were eligible to continue into the OLE Phase for up to 104 weeks of open-label avatrombopag therapy. Participants entering the OLE from the Core Study received a starting dose of open-label avatrombopag that was determined by the last dose of study drug at the End of Treatment (EOT) Visit (Visit 22) of the Core Study. Participants who discontinued the Core Study early because of lack of treatment effect and entered the OLE received open-label avatrombopag at a starting dose of 20 mg once daily of open-label avatrombopag.
Period: Core Study
Arm/Group | Eltrombopag (Core Study) | Avatrombopag (Core Study) | Avatrombopag (Open-label Extension Phase)
Started | 11 | 12 | 0
Completed | 0 | 1 | 0
Not Completed | 11 | 11 | 0
Not completed — Adverse Event, Non-Fatal | 0 | 1 | 0
Not completed — Lack of Efficacy | 5 | 1 | 0
Not completed — Study Terminated by Sponsor | 6 | 9 | 0
Period: Extension Phase
Arm/Group | Eltrombopag (Core Study) | Avatrombopag (Core Study) | Avatrombopag (Open-label Extension Phase)
Started | 0 | 0 | 6
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 6
Not completed — Adverse Event, Non-Fatal | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least one dose of study treatment and at least one postbaseline safety assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Eltrombopag (Core Study) | Avatrombopag (Core Study) | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Geometric Mean (Standard Deviation); unit: Years] | 45.4 (20.09) | 50.8 (23.04) | 48.2 (21.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Local Platelet Count for the 6 Month Treatment Period
Description: Platelet responses to avatrombopag was evaluated using the platelet counts determined at local clinical laboratories. Only participants with non-missing data at both baseline and the relevant post-baseline visit are included in the change from baseline summary statistics. Standard deviation is not applicable for some of the categories, from Visit 14 to Visit 22, as the number of participants analyzed for that visit was 1 individual.
Time Frame: Day 5, Day 8, Week 2, Week 3, Week 4, Week 6, Week 8, Week 10, Week 12, Week 14, Week 16, Week 18, Week 19, Week 20, Week 22, Week 23, Week 24, Week 25, Week 26
Population: The Full Analysis Set (FAS) included all participants who were randomized into the study. Only participants with non-missing data at both baseline and the relevant post-baseline visit are included in the change from baseline summary statistics.
Measure: Geometric Mean (Standard Deviation); unit: cells x 10^9/L
Arm/Group | Eltrombopag (Core Study) | Avatrombopag (Core Study)
Number analyzed (Participants) | 11 | 12
cells x 10^9/L
  Visit 3 (Day 5): number analyzed (Participants) | 10 | 10
  Visit 3 (Day 5) | 8.60 (17.312) | 12.85 (16.054)
  Visit 4 (Day 8): number analyzed (Participants) | 11 | 11
  Visit 4 (Day 8) | 32.50 (44.519) | 47.00 (59.690)
  Visit 5 (Week 2) | 73.41 (79.885) | 171.71 (201.736)
  Visit 6 (Week 3): number analyzed (Participants) | 10 | 12
  Visit 6 (Week 3) | 67.20 (95.536) | 114.21 (117.172)
  Visit 7 (Week 4): number analyzed (Participants) | 9 | 12
  Visit 7 (Week 4) | 28.72 (38.437) | 108.79 (217.036)
  Visit 8 (Week 6): number analyzed (Participants) | 7 | 11
  Visit 8 (Week 6) | 57.21 (57.718) | 150.68 (134.902)
  Visit 9 (Week 8): number analyzed (Participants) | 4 | 8
  Visit 9 (Week 8) | 67.25 (46.055) | 121.31 (149.040)
  Visit 10 (Week 10): number analyzed (Participants) | 3 | 6
  Visit 10 (Week 10) | 92.67 (34.649) | 126.25 (90.602)
  Visit 11 (Week 12): number analyzed (Participants) | 3 | 5
  Visit 11 (Week 12) | 87.33 (72.616) | 185.10 (115.841)
  Visit 12 (Week 14 ): number analyzed (Participants) | 3 | 4
  Visit 12 (Week 14 ) | 104.33 (77.114) | 159.38 (116.746)
  Visit 13 (Week 16): number analyzed (Participants) | 2 | 4
  Visit 13 (Week 16) | 47.75 (2.475) | 123.88 (124.474)
  Visit 14 (Week 18): number analyzed (Participants) | 1 | 2
  Visit 14 (Week 18) | 107.50 (NA) — Standard deviation is not applicable. | 46.50 (53.740)
  Visit 15 (Week 19): number analyzed (Participants) | 1 | 2
  Visit 15 (Week 19) | 13.50 (NA) — Standard deviation is not applicable. | 29.50 (22.627)
  Visit 16 (Week 20): number analyzed (Participants) | 0 | 1
  Visit 16 (Week 20) |  | 50.50 (NA) — Standard deviation is not applicable.
  Visit 18 (Week 22): number analyzed (Participants) | 0 | 1
  Visit 18 (Week 22) |  | 75.50 (NA) — Standard deviation is not applicable.
  Visit 19 (Week 23): number analyzed (Participants) | 0 | 1
  Visit 19 (Week 23) |  | 104.50 (NA) — Standard deviation is not applicable.
  Visit 20 (Week 24): number analyzed (Participants) | 0 | 1
  Visit 20 (Week 24) |  | 106.50 (NA) — Standard deviation is not applicable.
  Visit 21 (Week 25): number analyzed (Participants) | 0 | 1
  Visit 21 (Week 25) |  | 120.50 (NA) — Standard deviation is not applicable.
  Visit 22 (Week 26): number analyzed (Participants) | 0 | 1
  Visit 22 (Week 26) |  | 58.50 (NA) — Standard deviation is not applicable.

ADVERSE EVENTS:
Time Frame: Up to 34 Weeks in the Core Study (including Titration, Treatment, Dose Taper, and Follow-up for those that did not enter the Extension Phase) and up to 112 weeks in the Extension Phase (including Conversion, Maintenance, Dose Taper, and Follow-up).
Description: Treatment emergent adverse events were collected. Core Study Safety Analysis Set (SAS): All participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment. OLE SAS: All participants who received at least 1 dose of avatrombopag (either in the Core or Extension Phase) and had a postdose safety assessment.
Groups:
- Avatrombopag (Extension Phase): Participants who met the eligibility requirements for the Open-label Extension (OLE) Phase or who discontinued the Core Study early because of lack of treatment effect were eligible to continue into the OLE Phase for up to 104 weeks of open-label avatrombopag therapy. Participants entering the OLE from the Core Study received a starting dose of open-label avatrombopag that was determined by the last dose of study drug at the End of Treatment (EOT) Visit (Visit 22) of the Core Study. Participants who discontinued the Core Study early because of lack of treatment effect and entered the OLE received open-label avatrombopag at a starting dose of 20 mg once daily of open-label avatrombopag.
Arm/Group | Eltrombopag (Core Study) | Avatrombopag (Core Study) | Avatrombopag (Extension Phase)
Serious Adverse Events (participants affected / at risk) | 0/11 | 2/12 | 4/17
Other Adverse Events (participants affected / at risk) | 11/11 | 11/12 | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (Core Study) (N=11) | Avatrombopag (Core Study) (N=12) | Avatrombopag (Extension Phase) (N=17)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 1
Bronchitis Moraxella (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Thrombophlebitis Septic (Infections and infestations) | 0 | 1 | 1
Chronic lymphotic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (Core Study) (N=11) | Avatrombopag (Core Study) (N=12) | Avatrombopag (Extension Phase) (N=17)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 1
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 1
Abnormal Sensation in Eye (Eye disorders) | 0 | 1 | 1
Eye disorder (Eye disorders) | 0 | 1 | 1
Eye irritation (Eye disorders) | 0 | 1 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 1
Eye Swelling (Eye disorders) | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Glossodynia (Gastrointestinal disorders) | 1 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 3 | 3
Oral Mucosal blistering (Gastrointestinal disorders) | 1 | 0 | 1
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1
Fatigue (General disorders) | 5 | 1 | 5
Oedema peripheral (General disorders) | 1 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 1
Bronchitis moraxella (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 2 | 4
Oral candidiasis (Infections and infestations) | 0 | 1 | 1
Thrombophlebitis septic (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 2
Platelet count increased (Investigations) | 0 | 1 | 1
Weight increased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 3 | 4
Dysgeusia (Nervous system disorders) | 0 | 1 | 1
Head discomfort (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 3 | 3 | 5
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 2 | 2
Sinus headache (Nervous system disorders) | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 3 | 4
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 1
Menorrhagia (Reproductive system and breast disorders) | 2 | 1 | 1
Nipple Pain (Reproductive system and breast disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Raynaud's phenomenon (Vascular disorders) | 1 | 0 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Lymphocyte count increased (Investigations) | 1 | 0 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0
Discomfort (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Study was terminated early (during the Extension Phase) due to significant enrollment changes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other